CLINICAL TRIAL: NCT01688492
Title: A Phase 2 Study Combining Ipilimumab With Abiraterone Acetate Plus Prednisone in Chemotherapy and Immunotherapy-naïve Patients With Progressive Metastatic Castration-resistant Prostate Cancer
Brief Title: Combining Ipilimumab With Abiraterone Acetate Plus Prednisone in Chemotherapy and Immunotherapy-naïve Patients With Progressive Metastatic Castration-resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Northwestern University (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-120
Record Dates: First submitted 2012-09-14; First posted 2012-09-20 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: MDX-010 (Ipilimumab); ABIRATERONE ACETATE (CB 7630); PREDNISONE; Immunotherapy-naïve; castration resistant prostate cancer (CRPC); 12-120
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab

ARMS (1):
- ipilimumab (Experimental): This multi-institution open label study has a Phase 1 and Phase 2 component. The Phase 1 dose escalation stage is to establish the tolerability of ipilimumab to be used in combination with the standard clinical dose of abiraterone acetate plus prednisone in chemotherapy and immunotherapy-naïve patients with progressive metastatic CRPC. Due to the overlapping potential hepatic toxicity between abiraterone and ipilimumab, a Lead in Therapy with abiraterone plus prednisone for 2 cycles will assess for adverse events related to the abiraterone plus prednisone. Patients, who tolerate well the Lead in therapy as defined by Grade 1 or less AEs, will pursue Combination Therapy. Patients with AEs Grade ≥ 2 after Lead in Therapy will be excluded and replaced. The Phase 2 stage will assess efficacy and confirm an acceptable safety profile of the recommended dose.
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Abiraterone acetate (JanssenBiotech, Inc/Johnson & Johnson) 1000 mg orally daily plus prednisone 5 mg orally twice daily will be administered continuously during the duration of the trial. Starting at cycle 3 (Combination Therapy), Ipilimumab (Bristol-Myers Squibb) will be infused intravenously (IV) once every 3 weeks for a total of 4 infusions.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, taking ipilimumab with abiraterone acetate plus prednisone has on the patient and the prostate cancer. Abiraterone acetate plus prednisone are drugs that lower testosterone (testosterone stimulates prostate cancer growth). Abiraterone acetate plus prednisone is a treatment for patients with prostate cancer.

Abiraterone acetate plus prednisone has not been used together with ipilimumab before. This study will test how they work together. Each patient will receive abiraterone acetate, prednisone and ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

Chemotherapy- and immunotherapy-naïve patients with progressive metastatic CRPC are eligible.

* Age 18 or older, and be willing and able to provide informed consent.
* Histologically or cytologically confirmed adenocarcinoma of the prostate at either MSKCC or at the participating site.
* Castrate serum testosterone level, ≤ 1.73 nmol/L (50 ng/dL), at the Screening visit.
* Ongoing androgen deprivation therapy with a GnRH analogue or bilateral orchiectomy (ie, surgical or medical castration).
* Metastatic disease on imaging (e.g., bone scan, CT, MRI). Patients whose disease spread is limited to regional pelvic lymph nodes are not eligible. If lymph node metastasis is the only evidence of metastasis, it must be ≥ 2 cm in diameter.
* Progressive disease at study entry defined by PSA and/or radiographic criteria according to the PCWG2.
* Karnofsky performance status of ≥80-100, and estimated life expectancy of ≥ 6 months.
* Toxicities related to prior therapy must either have returned to ≤ Grade 1 or baseline or been deemed irreversible and in the opinion of the Investigator not worsened.
* Able to swallow the study drug and comply with study requirements.

Exclusion Criteria:

* History of another malignancy within the previous 5 years other than nonmelanomatous skin cancer.
* Absolute neutrophil count < 1,500/μL, or platelet count < 75,000/μL, or hemoglobin < 5.6 mmol/L (9 g/dL) at the Screening visit. (NOTE: patients may not have received any growth factors within 7 days or blood transfusions within 28 days of the hematologic laboratory values obtained at the Screening visit).
* Serum bilirubin ≥ 1.5 x ULN or for patients with Gilbert's disease, ≥3 mg/dL at the Screening visit; AST or ALT ≥ 2.5 x ULN, (for patients with known liver metastasis, AST or ALT ≤ 5 x ULN is allowed) at the Screening visit.
* Creatinine > 177 μmol/L (2 mg/dL), albumin < 30 g/L (3.0 g/dL), potassium ≤ 3.5 mEq/L at the Screening visit.
* Clinically significant cardiovascular disease including myocardial infarction within 6 months, uncontrolled angina within 3 months, congestive heart failure New York Heart Association (NYHA) class 3 or 4, uncontrolled hypertension as indicated by systolic blood pressure > 160 mmHg or diastolic blood pressure > 95 mmHg at the Screening visit.
* Major surgery or radiation therapy within 4 weeks of enrollment (Day 1 Visit).
* Treatment with antiandrogens (eg, bicalutamide, flutamide, or nilutamide) within 4 weeks of enrollment (Day 1 visit). Concomitant therapy with any of the agents listed in Section 4.3.2 is prohibited.
* History of progression of prostate cancer disease while receiving ketoconazole. Prior use or participation in a clinical trial of an investigational agent that blocks androgen synthesis (eg, abiraterone acetate, TAK-700, TAK-683, TAK-448), chemotherapy, or immunological agents (eg, immune modulators, cytokines, vaccines, or antibody-delivered chemotherapy). The use of denosumab for bone metastasis is permitted.
* Known allergy to any of the compounds under investigation.
* The patient has uncontrolled or significant medical condition other than cancer, that would prevent the participation in the study or make this protocol unreasonably hazardous, in the opinion of the investigator, including but not limited to:
* Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's granulomatosis]); motor neuropathy considered of autoimmune origin (eg, Guillain-Barre syndrome and myasthenia gravis).
* Known or suspected brain metastasis, or untreated leptomeningeal disease.
* Active infection or other medical condition that would make prednisone use contraindicated.
* Active or symptomatic viral hepatitis or chronic liver disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2012-09; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
safety (Phase I) | 2 years
  AEs will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grading scale, version 4.0.
progression-free survival (PFS) Phase II | 8 months
  which is defined as the time from the start of therapy until the criteria for progression are met

SECONDARY OUTCOMES:
Changes in PSA kinetics | 2 years
  PSA levels will be assessed every 4 weeks during the Lead in Therapy, every 3 weeks during the Combination Therapy and every 4 weeks during the Maintenance Therapy. Outcomes will be reported both by the percent change in PSA from baseline and Week 21 (or earlier for those who discontinue therapy) and the maximum decline in PSA using a waterfall plot.
Measurable disease when present | 2 years
  Measurable disease in viscera (liver or lung) is defined as per PCWG2 modified RECIST 1.1 as a lesion ≥10 mm in its longest diameter as measured with conventional techniques (ie, CT or MRI). For a lymph node to be considered measurable, the minimum diameter must be ≥20 mm in long axis when assessed by CT scan. All other lesions (or sites of disease) will be considered nonmeasurable disease.
Evaluate changes in radionuclide bone scan | 2 years
  Radionucleotide bone scan outcome should be recorded as either new lesions or no new lesions. On bone scan, progression of bone metastases is defined as the appearance of 2 or more new bone lesions compared to the baseline scan. In the case of the first Week 8 and Week 16 assessment scans a confirmatory scan performed 6 weeks later needs to shows 2 or more additional new lesions (for a total of at least 4 new lesions seen since baseline) for progression to be documented (the date of progression is always the date of the first scan showing the change).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Danila, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Northwestern University, Evanston, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/